CLINICAL TRIAL: NCT05560308
Title: A Prospective, Multicenter，Phase II Clinical Study of Trastuzumab and Pyrotinib Maleate in Patients With HER2-positive Metastatic Breast Cancer Who Had Progressed on TKI Therapy
Brief Title: Phase II Clinical Study of T-DM1 and Pyrotinib Maleate in Patients With HER2-positive Metastatic Breast Cancer Who Had Progressed on TKI Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC- T-DM1
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: HER2+ Advanced Breast Cancer Patients Progressing on TKI Therapy
MeSH Terms: interventions — Ado-Trastuzumab Emtansine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trastuzumab Emtansine for Injection；Pyrotinib Maleate Tablets (Experimental): Trastuzumab Emtansine for Injection: 3.6 mg/kg body weight (IV), administered on day 1, 21 days as a treatment cycle; Pyrotinib Maleate Tablets: The initial dose is 320 mg (PO), administered orally within 30 minutes after meals, at the same time every day, 21 days as a treatment cycle; Efficacy was assessed every two cycles and treatment was continued until disease progression or intolerable toxicity or death.
  Interventions: Drug: Trastuzumab Emtansine for Injection; Drug: Pyrotinib Maleate Tablets

INTERVENTIONS:
Drug: Trastuzumab Emtansine for Injection — 3.6 mg/kg body weight (IV), administered on day 1, 21 days as a treatment cycle;
Drug: Pyrotinib Maleate Tablets — The initial dose is 320 mg (PO), administered orally within 30 minutes after meals, at the same time every day, 21 days as a treatment cycle;

SUMMARY:
This trial is a combination of trastuzumab and pyrotinib in the treatment of patients with HER2-positive metastatic breast cancer who have progressed on TKI therapy. A total of 50 patients were enrolled in the study design. Preliminary efficacy and safety in patients with HER2-positive metastatic breast cancer who have progressed on TKI therapy.

ELIGIBILITY:
Inclusion criteria：

1. Female breast cancer patients aged ≥18 years and ≤75 years old
2. HER2 positive (IHC3+, or IHC2+ and positive FISH test) confirmed by the center
3. ECOG score 0-1
4. Patients with advanced breast cancer who have progressed on lapatinib or pyrotinib
5. There are measurable lesions
6. Left ventricular ejection fraction (LVEF) ≥ 50%
7. 12-lead ECG: Fridericia-corrected QT interval (QTcF) in women < 470 ms;
8. The function level of major organs must meet the following requirements: blood routine: ANC≥1.5×109/L; PLT≥90×109/L; Hb≥90g/L; blood biochemistry: TBIL≤2.5×ULN; ALT and AST≤2.5 ×ULN; BUN and Cr ≤ 1.5×ULN;
9. For female subjects who are not menopausal or surgically sterilized, agree to abstain from sex or use effective contraceptive methods during the treatment period and for at least 2 months after the last dose in the study treatment;
10. Voluntarily join the study, sign informed consent, have good compliance and be willing to cooperate with follow-up.

exclusion criteria：

1. Patients who have previously used ADCs to treat advanced breast cancer
2. Symptomatic patients with brain metastases
3. Control unstable pleural effusion and ascites patients
4. Patients with previous or concurrent malignancies whose natural medical history or treatment may interfere with the safety or efficacy assessment of the study protocol are not eligible to participate in this trial, except for basal cell or squamous cell skin cancer, cervical cancer in situ, or bladder cancer , or the subject has lived free of disease (other cancers) for at least 5 years.
5. Active infection requiring systemic treatment
6. Gastrointestinal dysfunction or disease that may seriously affect the absorption of the study drug (such as ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) or severely impair the ability to swallow capsules/tablets
7. Known history of myelodysplastic syndrome or acute myeloid leukemia
8. History of abdominal fistula, gastrointestinal perforation or abdominal abscess within 28 days
9. Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months
10. History of acute coronary syndrome (including myocardial infarction, unstable angina, coronary artery, arterial bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 6 years
11. Symptomatic congestive heart failure (New York Heart Association III-IV) or cardiomyopathy with left ventricular ejection fraction (LVEF) <50%
12. Clinically significant ventricular arrhythmia (sustained tachycardia/ventricular fibrillation) or high-grade AV block (eg, bifascicular block, Mobitz type II, and third-degree AV block), unless fitted pacemaker
13. Any concurrent severe and/or uncontrolled medical conditions that, in the judgment of the investigator, would result in unacceptable safety risks, prohibit subjects from participating in clinical studies, or affect protocol compliance

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with advanced breast cancer aged ≥18 years and ≤75 years old
Enrollment: 50 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-08-23 (Estimated)

PRIMARY OUTCOMES:
ORR(objective response rate) | Estimated 24 months
  rate of CR and PR in all subjects